CLINICAL TRIAL: NCT07376902
Title: Effects of White Noise on Academic Skills in Children With ADHD and Specific Learning Disorders: New Perspectives for Personalised Rehabilitation and Educational Intervention
Brief Title: White Noise in SLD and ADHD
Acronym: WHITE NOISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 137/SR/24
Record Dates: First submitted 2025-12-17; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; Specific Learning Disorder; Specific Learning Disability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Specific Learning Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD (Experimental): Subjects are enrolled according to the following criteria: Intelligence Quotient (IQ), assessed using the Wechsler Intelligence Scales (WISC-IV), ≥ 70. Age between 8 and 13 years. Diagnosis of ADHD according to DSM-5 criteria.
  Interventions: Other: White noise; Other: No white noise
- ADHD + SLD (Experimental): Subjects are enrolled according the following criteria: Intelligence Quotient (IQ), assessed using the Wechsler Intelligence Scales (WISC-IV), ≥ 70. Age between 8 and 13 years. Diagnosis of SLD with comorbid ADHD according to DSM-5 criteria.
  Interventions: Other: White noise; Other: No white noise

INTERVENTIONS:
Other: White noise — Reading and writing standardized assessment with white noise. The white noise, created for this study by an audio engineer, is played through a speaker positioned approximately 1 m from the participant, at an intensity of 60-65 dB within the designated testing environment. At the start of each session, participants are informed of its presence to prevent any potential discomfort. This adaptation phase lasts approximately 2-3 minutes.
Other: No white noise — Reading and writing standardized assessment in the absence of white noise.

SUMMARY:
White noise has been shown to improve working memory and attention in children diagnosed with ADHD . These cognitive abilities are fundamental to the acquisition of reading and writing skills. Therefore, the aim of the present study is to evaluate the effects of white noise on reading and writing performance in children with a diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD) and Specific Learning Disorder (SLD) attending the first and second cycles of primary school.

The study is a randomized crossover clinical trial comprising five sequential phases. Each participant completes two standardized assessment sessions, one with white noise and one without, in a randomized order, separated by a four-week interval.

* Phase I (Recruitment and Screening): potential participants are identified and assessed for eligibility at the Centro di Riabilitazione San Raffaele Pisana in Rome.
* Phase II (Diagnostic Grouping): eligible children are assigned to one of two diagnostic groups based on their clinical profile (Group SLD + ADHD or Group SLD-only).
* Phase III (Randomized Sequencing): Within each diagnostic group, participants are randomly allocated to one of two exposure sequences to counterbalance order effects (White-noise → No-noise, or No-noise → White-noise).
* Phase IV (First Assessment Session): standardized assessment under randomized conditions, with or without white noise.
* Phase V (Second Assessment Session): standardized assessment, conducted four weeks later, with or without white noise according to the previous randomization.

ELIGIBILITY:
Inclusion Criteria:

* Intelligence Quotient (IQ), assessed using the Wechsler Intelligence Scales (WISC-IV), ≥ 70.
* Age between 8 and 13 years.
* Diagnosis of SLD, with or without comorbid ADHD according to DSM-5 criteria.

Exclusion Criteria:

* Genetic disorders or sensory deficits.
* Pharmacological treatments that could interfere with task performance (including methylphenidate or specific ADHD treatments).

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Reading speed | 4 weeks
  For the passage-reading test and the word- and nonword-reading tasks: reading speed, expressed in syllables per second (syl/sec) was calculated by dividing the total number of syllables in the stimulus by the total reading time, measured in seconds.
Reading Accuracy | 4 weeks
  For the passage-reading test and the word- and nonword-reading tasks reading accuracy was defined as the total number of errors produced.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No